CLINICAL TRIAL: NCT07143019
Title: p48/64 MW HPC in Aneurysm Occlusion (PIANO): Prospective, Multicenter, Single-arm Clinical Trial to Determine Safety and Effectiveness of the Flow Modulation Device in the Treatment of Wide-necked Intracranial Aneurysms.
Brief Title: The Use of p48/64 MW HPC Flow Modulation Device in the Treatment of Wide-necked Intracranial Aneurysms
Acronym: PIANO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: phenox Inc. (Industry)
Collaborators: Phenox GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCT-002-23
Record Dates: First submitted 2025-08-12; First posted 2025-08-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hemorrhagic Stroke; Aneurysm, Intracranial; Saccular Aneurysm; Fusiform Aneurysm; Brain Aneurysm
Keywords: Neurovascular Intervention; phenox; Brain; Unruptured Aneurysm; Flow diversion; Flow diverter; Occlusion; Flow modulation device
MeSH Terms: conditions — Hemorrhagic Stroke; Intracranial Aneurysm; Aneurysm; Bites and Stings

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, single-arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Intervention/Treatment (Experimental): Device: Flow diversion using the p48 MW HPC Device: Flow diversion using the p64 MW HPC
  Interventions: Device: Flow diversion

INTERVENTIONS:
Device: Flow diversion — The p48 MW HPC and p64 MW HPC flow modulation device is indicated for use in the treatment of intracranial aneurysms (IAs) arising from a parent vessel with a diameter of ≥2.0mm and ≤5.0 mm.

SUMMARY:
To determine safety and effectiveness of the p48 MW HPC and p64 MW HPC flow diverter in the treatment of wide-necked intracranial aneurysms.

DETAILED DESCRIPTION:
To assess safety, effectiveness, and performance of the p48/p64 MW HPC flow diverter in the endovascular treatment of wide-necked intracranial aneurysms (IA) at 12 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years
2. Subject has a mRS ≤2 before the index procedure
3. Subject has an unruptured or recanalized intracranial aneurysm (IA). The subject may also have a previous ruptured aneurysm, provided rupture of this aneurysm has occurred more than 30 days from the index procedure. The IA must have the following characteristics below:

   1. Saccular or fusiform morphology
   2. Located in the internal carotid artery and its branches
   3. Aneurysm neck ≥4 mm or dome-to-neck ratio <2
   4. Parent vessel diameter ≥2.0mm and ≤5.0mm both distal and proximal to the target IA
4. Subject or subject's legally authorized representative (LAR) has provided written informed consent and has agreed to comply with study procedures.

Exclusion Criteria:

1. Previous flow diverter or stent within the parent vessel of the target aneurysm to be treated
2. Any other known IA requiring treatment within 3 months post-procedure
3. Subarachnoid hemorrhage in the past 30 days prior to the index procedure
4. Has a true bifurcation aneurysm, defined as an aneurysm (saccular or non-saccular) located at the point of vessel bifurcation
5. Anatomy unsuitable for endovascular procedure due to severe vessel tortuosity or stenosis, or stented ipsilateral carotid artery within 3 months prior to the index procedure
6. Subject with a brain arteriovenous malformation (AVM) or other vascular malformation in the area of the target aneurysm
7. Major surgery in the last 30 days, including endovascular procedures, or is planned in the next 90 days after enrollment date
8. Unstable neurologic deficit (i.e., any worsening of clinical condition in the last 30 days)
9. Known serious sensitivity to radiographic contrast agents that cannot be managed medically
10. Known sensitivity to nickel, titanium metals or their alloys or any other investigational device components
11. Irreversible bleeding disorder and/or signs of active bleeding at subject presentation
12. Known renal failure with a serum creatinine >2.5 mg/dl (or 220 μmol/l) not on dialysis
13. Contraindication to CT scan, MRI, or angiography
14. Contraindication or known allergies to anticoagulants or antiplatelets (e.g. aspirin, heparin, clopidogrel, prasugrel, or ticagrelor)
15. Known coagulopathy, or an admission International Normalized Ratio >3.0 without oral anticoagulation therapy, or an admission platelet count of <100000
16. Has acute life-threatening illness other than the neurological disease (i.e., acute kidney or heart failure) to be treated in this trial
17. Unable to complete the required study follow-ups
18. Evidence of active infection at the time of treatment (e.g., fever, elevated white blood cell count)
19. Participating in another clinical trial that could affect participation or primary outcomes of this study
20. Women currently pregnant or wish to become pregnant during the study or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy and Performance Endpoint: Number of subjects with 100% occlusion of the target aneurysm without significant parent artery stenosis and no retreatment of the target aneurysm from the index procedure to the 12-month follow-up visit. | 12 months
  The Primary Efficacy and Performance Endpoint is a composite of 100% target aneurysm occlusion (Raymond-Roy Class I) without significant stenosis (defined as ≤50% stenosis) of the parent artery based on independent core lab evaluation of the 12-month follow-up angiogram (DSA), and no subsequent treatment at the target aneurysm at the 12-month follow-up visit.
The Primary Safety Endpoint: Number of subjects with ischemic or hemorrhagic stroke or neurologic death from treatment to 12-months, as adjudicated by a Clinical Events Committee. | From treatment - 12 months
  The Primary Safety Endpoint is the incidence of major stroke (ischemic or hemorrhagic) in the territory supplied by the treated artery, defined as an increase in NIHSS score by 4 points, or neurologic death within 1 year after treatment.

SECONDARY OUTCOMES:
Secondary Safety Endpoint #1: Number of subjects with a modified Rankin Scale (mRS) score > 2 | 30 days post procedure and at the following timepoints: 6-month, 1 year, 3 years, and 5 years
  Morbi-mortality refers to the combined study of morbidity (the state of being diseased or unhealthy) and mortality (the state of being subject to death) that results in a modified Rankin Scale (mRS) score > 2
Secondary Safety Endpoint #2: Number of subjects with procedural and/or device-related serious adverse events (SAE) | 30 days post procedure and at the following timepoints: 6-months, 1 year, 3 years, and 5 years
  The number of subjects that have a reported event related to the procedure, the device (based on FDAs definition of a serious adverse event), or both will be analyzed by an independent Clinical Events Committee
Secondary Safety Endpoint #3: Number of subjects with a neurologic event of interest defined as any death, neurological death, target aneurysm rupture or re-rupture, target aneurysm retreatment, or intracranial hemorrhage | 30 days post procedure and at the following timepoints: 6-months and 12-months post procedure
  The number of subjects who have died by any cause, who have had their treated target aneurysm rupture or re-rupture, who have had their target aneurysm retreated, or who have had an intracranial hemorrhage, as adjudicated by an independent Clinical Events Committee

OTHER OUTCOMES:
Additional Analysis #1: Number of subjects with 100% occlusion (Raymond-Roy Class I) of the target aneurysm at follow-up visits | Post procedure: 6-months, 1 year, 3 years and at 5 years
  The number of subjects with 100% occlusion (Raymond-Roy Class I) of the target aneurysm at follow-up visits will be analyzed
Additional Analysis #2: Number of subjects with retreatment of the target aneurysm | Post Procedure: 6-months, 1 year, 3 years, and at 5 years
  The number of subjects with target aneurysm retreatment will be analyzed
Additional Analysis #3: Number of subjects with a target aneurysm recanalization/recurrence | Post procedure: 6-months, 1 year, 3 years, and at 5 years
  The number of subjects with target aneurysm recanalization or recurrence will be analyzed
Additional Analysis #4: Number of subjects with significant (> 50% stenosis) parent artery stenosis, as assessed independent core laboratory post-procedure | Post procedure: 6-months, 1 year, 3 years, and at 5 years
  The number of subjects with significant (> 50% stenosis) parent artery stenosis, as assessed post-procedure by independent core lab will be analyzed
Additional Analysis #5: Number of subjects with technical device success defined as complete coverage of the target aneurysm with ≥1 FMD) per subject at the target site during the index procedure | Immediately after the Index Procedure
  The number of subjects with complete coverage of the target aneurysm with ≥1 FMD per subject at the target site during the index procedure, as assessed by the independent core lab

CONTACTS AND LOCATIONS:
Overall Officials: Demetrius Lopes, MD, Principal Investigator — Advocate Aurora Research Institute, LLC; Jared Knopman, MD, Principal Investigator — The Joan and Sanford I. Weill Medical College of Cornell University; Eytan Raz, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Baptist Health Research Institute, Jacksonville, Florida
  - UBNS, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No